CLINICAL TRIAL: NCT00315211
Title: Phase 2 Study of Weekly Topotecan With Docetaxel for Recurrent Small Cell Lung Cancer
Brief Title: Weekly Topotecan With Docetaxel in Recurrent Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Aultman Health Foundation (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hycamtin study #102143; Lung 01 (Other: Aultman Health Foundation)
Record Dates: First submitted 2006-04-17; First posted 2006-04-18 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Mediastinal Neoplasms
Keywords: Small Cell Lung Cancer Recurrent
MeSH Terms: conditions — Mediastinal Neoplasms | interventions — Topotecan; Docetaxel

ARMS (1):
- Arm A (Other): Weekly intravenous topotecan with intravenous docetaxel
  Interventions: Drug: Intravenous Topotecan; Drug: Intravenous Docetaxel

INTERVENTIONS:
Drug: Intravenous Topotecan — Topotecan 3 mg/m2 IV over 30 minutes on Days 1 and 8 every 21 days
  Other Names: Hycamtin
Drug: Intravenous Docetaxel — Docetaxel 30 mg/m2 IV over 60 minutes on Days 1 & 8 of a 21 day cycle
  Other Names: Taxotere

SUMMARY:
The purposes of this study are:

* To determine the overall response rate of patients treated with at least 2 cycles of this regimen.
* To determine the feasibility and toxicity of the combination of topotecan and docetaxel.

DETAILED DESCRIPTION:
The main objective of this study was to determine the overall response rate of patients treated with at least 2 cycles of topotecan and docetaxel. The secondary objectives were to determine the feasibility and toxicities of this combination. The final secondary objective is overall survival for patients that received 2 or more cycles.

Methods: Eligible pts with recurrent small cell lung cancer had to be at least 3 months from initial treatment. Pts received Docetaxel 30 mg/m2 IV followed by Topotecan 3 mg/m2 IV Days 1 and 8 of a 21 day cycle. Disease assessment was done every 2 cycles. Toxicity was measured each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Recurred greater than 90 days after initial treatment
* At least 1 measurable lesion
* Only 1 prior chemotherapy
* Must be over 18 years of age
* ECOG performance status of 0 - 2
* Adequate hematologic, renal, and hepatic function

Exclusion Criteria:

* No prior use of topotecan, docetaxel, or irinotecan
* No symptomatic brain metastases
* History of cardiac arrhythmias, congestive heart failure, stroke, or embolic events
* No prior investigational agents within 1 month prior
* Lung cancer of mixed histology
* Known uncontrolled seizure disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-11; Primary Completion 2007-06 (Actual); Study Completion 2007-11-08 (Actual)

PRIMARY OUTCOMES:
To determine the overall response rate of patients treated with at least two cycles of topotecan and docetaxel | 3 years
  To determine the overall response rate of patients treated with at least two cycles of topotecan and docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: Raza Khan, MD, Principal Investigator — Aultman Hospital
Locations (1):
- Aultman Hospital, Canton, Ohio, United States